CLINICAL TRIAL: NCT02634645
Title: A Multicenter Prospective Study Evaluating Outcomes of Endoscopic Eradication Therapy in Patients With Barrett's Esophagus Associated Neoplasia: The TREAT-BE (Treatment With Resection and Endoscopic Ablation Techniques for Barrett's Esophagus) Consortium
Brief Title: TREAT-BE Study (Treatment With Resection and Endoscopic Ablation Techniques for Barrett's Esophagus)
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Northwestern University Feinberg School of Medicine (Other); University of California, Los Angeles (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); California Pacific Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14-2371
Record Dates: First submitted 2015-06-08; First posted 2015-12-18 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Barrett's Esophagus; Esophageal Cancer
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms | interventions — Esophagectomy; Drug Therapy; Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Barrett's Esophagus: Patients with non-dysplastic Barrett's esophagus, patients with Barrett's related dysplasia which includes low-grade dysplasia, high-grade dysplasia and intramucosal cancer who will be evaluated and treated with endoscopic eradication therapies (EET).
  Interventions: Procedure: Endoscopic eradication therapies (EET)
- Patients with invasive esophageal cancer: Patients with invasive esophageal cancer who will be treated with surgery (esophagectomy), chemotherapy, radiation, and palliative treatment modalities.
  Interventions: Procedure: Esophagectomy; Drug: Chemotherapy; Radiation: Radiation

INTERVENTIONS:
Procedure: Endoscopic eradication therapies (EET) — Endoscopic eradication therapies (EET) includes endoscopic mucosal resection (EMR), which describes the process by which the area most likely to harbor highest grade of dysplasia/neoplasia is removed; radiofrequency ablation (RFA), which describes the process by which Barrett's segments are removed via burning/ablation; and cryotherapy.
  Groups: Patients with Barrett's Esophagus
Procedure: Esophagectomy — The esophagus is surgically removed
  Groups: Patients with invasive esophageal cancer
Drug: Chemotherapy — Chemical substances are used to treat cancer
  Groups: Patients with invasive esophageal cancer
Radiation: Radiation — Cancer cells are destroyed by radiation therapy.
  Groups: Patients with invasive esophageal cancer

SUMMARY:
A prospective outcomes study in patients with and esophageal cancer (EAC) and Barrett's esophagus (BE) associated neoplasia being evaluated for endoscopic eradication therapy (EET).

DETAILED DESCRIPTION:
Patients will be enrolled in this study at the participating centers when evaluated in gastro-intestinal (GI) clinics and endoscopy suites. Initial evaluation of patients will include collection of data on demographics, assessment of risk factors such as smoking, metabolic syndrome, family history and detailed medication history, and past surgical history. All patients will be complete questionnaires regarding Gastroesophageal Reflux Disease (GERD) symptoms, GERD related quality of life (QOL) and overall health related QOL. Details of all previous endoscopic and surgical evaluation along with histopathology data will be documented. Patients undergoing endoscopic evaluation at the participating centers will have their endoscopic and histopathology results documented. This will include data collection regarding use of advanced imaging techniques, details regarding tissue acquisition, EET and adverse events. Patients undergoing esophagectomy will have surgical details documented along with complications related to surgery. Similarly, details regarding chemoradiation treatments will be documented .

ELIGIBILITY:
Inclusion Criteria:

* Patients with Barrett's related neoplasia and dysplasia. Patients with esophageal cancer

Exclusion Criteria:

* Patients with squamous cell carcinoma

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Formation of a multi-site prospective database of patients with BE associated neoplasia referred for consideration for EET and EAC.
  Women and minorities will be included as they are found to have BE, BE related dysplasia, and EAC. It is well recognized that the majority of patients diagnosed with BE are white males. However, we will actively seek to include all women and minorities with a diagnosis of BE associated neoplasia for the study.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-01; Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Overall improvement of patient outcomes in patients treated with endoscopic eradication therapy (EET). | 5 years
  A systematic, prospective collection of data from a large cohort of patients with BE and EAC undergoing EET will provide useful data in effort to improve overall patient outcomes.

SECONDARY OUTCOMES:
Long-term effectiveness or durability of EET in BE related neoplasia. | 5 years
  To report on long-term effectiveness or durability of EET in BE related neoplasia.
Quality of life (QOL) in patients undergoing endoscopic eradication therapies for Barrett's associated neoplasia | 5 years
  To assess quality of life (QOL) using the Promise GERD HRQL (Health Related Quality of Life) questionnaire in patients undergoing endoscopic eradication therapies for Barrett's associated neoplasia
Recurrence rate of neoplasia | 5 years
  To report on the recurrence rate of neoplasia (defined as number of patients with established eradicated neoplasia post-EET who are found to have recurrent intestinal metaplasia on subsequent surveillance biopsies)
Recurrence rate of intestinal metaplasia | 5 years
  To report on the recurrence rate intestinal metaplasia (defined as number of patients with established eradicated intestinal metaplasia and/or neoplasia post-EET who are found to have recurrent intestinal metaplasia on subsequent surveillance biopsies).
Recurrence rate based on baseline dysplasia, Barrett's length, and treatment modality | 5 years
  Percentage of patients of different baseline Barrett's treatment modalities (EMR vs. RFA vs. cryotherapy) whose Barrett's is persistent despite treatment and/or recurs post-eradication. Percentage of patients of different baseline Barrett's lengths whose Barrett's is persistent despite treatment and/or recurs post-eradication. Percentage of patients of different baseline Barrett's histologies (i.e. high grade dysplasia/intramucosal cancer vs. low grade dysplasia) whose Barrett's is persistent despite treatment and/or recurs post-eradication.
Persistence rate based on baseline dysplasia, Barrett's length, and treatment modality | 5 years
  Percentage of patients of different baseline Barrett's treatment modalities (EMR vs. RFA vs. cryotherapy) whose Barrett's is persistent despite treatment and/or recurs post-eradication. Percentage of patients of different baseline Barrett's lengths whose Barrett's is persistent despite treatment and/or recurs post-eradication. Percentage of patients of different baseline Barrett's histologies (i.e. high grade dysplasia/intramucosal cancer vs. low grade dysplasia) whose Barrett's is persistent despite treatment and/or recurs post-eradication.
Adverse event rates associated with EET for BE associated neoplasia and EAC. | 5 years
  To determine adverse event rates associated with EET for BE associated neoplasia and EAC.
Determine health-care utilization including endoscopic surveillance practices and outcomes in BE patients with and without neoplasia | 5 years
  Number of BE patients (both with and without neoplasia) in the general population who receive various endoscopic interventions (including RFA, cryotherapy, EMR, endoscopic surveillance)
Magnitude of risk factors for BE. | 5 years
  The number of BE patients who fall into specific age cohorts; the number of BE patients who are male/female; the number of BE patients who fall into specific BMI cohorts; the number of BE patients who have used tobacco and/or currently use tobacco; the number of BE patients who have GERD symptoms; the number of BE patients who have metabolic syndrome; the number of BE patients who take aspirin, NSAIDS, anti-hyperglycemic medications, and/or statins.
Magnitude of risk factors for BE related neoplasia. | 5 years
  The number of BE related neoplasia patients who fall into specific age cohorts; the number of BE related neoplasia patients who are male/female; the number of BE related neoplasia patients who fall into specific BMI cohorts; the number of BE related neoplasia patients who have used tobacco and/or currently use tobacco; the number of BE related neoplasia patients who have GERD symptoms; the number of BE related neoplasia patients who have metabolic syndrome; the number of BE related neoplasia patients who take aspirin, NSAIDS, anti-hyperglycemic medications, and/or statins.
Magnitude of risk factors for EAC. | 5 years
  The number of EAC patients who fall into specific age cohorts; the number of EAC patients who are male/female; the number of EAC patients who fall into specific BMI cohorts; the number of EAC patients who have used tobacco and/or currently use tobacco; the number of EAC patients who have GERD symptoms; the number of EAC patients who have metabolic syndrome; the number of EAC patients who take aspirin, NSAIDS, anti-hyperglycemic medications, and/or statins.
Impact of endoscopic and radiologic imaging modalities. | 5 years
  Number of patients whose treatment plan changes due to endoscopic ultrasound and/or Computed Tomography-Positron Emission Tomography (CT-PET) findings
Median time to recurrence of intestinal metaplasia | 5 years
  To report on the median time to recurrence (measured median amount of months between complete eradication and recurrence of intestinal metaplasia).
Median time to recurrence of neoplasia | 5 years
  To report on the median time to recurrence (measured median amount of months between complete eradication and recurrence of neoplasia).

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Wani, MD, Principal Investigator — University of Colorado, Denver
Locations (4):
- United States (4):
  - UCLA Medical Center, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Washington University, St Louis, Missouri

REFERENCES:
- [Derived] Wani S, Han S, Kushnir V, Early D, Mullady D, Hammad H, Brauer B, Thaker A, Simon V, Ezekwe E, Hollander T, Wood M, Rastogi A, Edmundowicz S, Muthusamy VR, Komanduri S. Recurrence Is Rare Following Complete Eradication of Intestinal Metaplasia in Patients With Barrett's Esophagus and Peaks at 18 Months. Clin Gastroenterol Hepatol. 2020 Oct;18(11):2609-2617.e2. doi: 10.1016/j.cgh.2020.01.019. Epub 2020 Jan 23. PMID 31982610
- [Derived] Omar M, Thaker AM, Wani S, Simon V, Ezekwe E, Boniface M, Edmundowicz S, Obuch J, Cinnor B, Brauer BC, Wood M, Early DS, Lang GD, Mullady D, Hollander T, Kushnir V, Komanduri S, Muthusamy VR. Anatomic location of Barrett's esophagus recurrence after endoscopic eradication therapy: development of a simplified surveillance biopsy strategy. Gastrointest Endosc. 2019 Sep;90(3):395-403. doi: 10.1016/j.gie.2019.04.216. Epub 2019 Apr 17. PMID 31004598